CLINICAL TRIAL: NCT05296187
Title: Efficacy of Transcutaneous Electrical Acupuncture Point Stimulation (TEAS) for the Prevention of Propofol Injection Pain in Children
Brief Title: Efficacy of TEAS On Prevention of Propofol Injection Pain in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TEAS Propofol Injection Pain
Record Dates: First submitted 2022-03-14; First posted 2022-03-25 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Injection Site

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP TEAS (Active Comparator): Patients will receive TEAS bilaterally at two acupoints: Hegu (L14) and Neiguan (PC6).
  Interventions: Device: TEAS
- Control Sham Group (Placebo Comparator): Patients in the sham group will be undergoing electrode attachment on the target acupoints without electronic stimulation.
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS — Transcutaneous electrical acupuncture stimulation

SUMMARY:
The purpose of this study is to determine the efficacy of transcutaneous electrical acupoint stimulation for the prevention of propofol injection pain in children.

DETAILED DESCRIPTION:
Pain from the injection of propofol is a common side effect during anesthetic practice. Various methods have been used to reduce this pain. This prospective, randomized study was designed to determine the efficacy of transcutaneous electrical acupuncture point stimulation in reducing propofol injection pain in children.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II and aged 6-13 years patents who will undergo elective surgery under general anesthesia

Exclusion Criteria:

* patients with propofol allergy
* patients who have renal, hepatic, cardiac, neurological, psychiatric disease
* Cardiac and cranial surgery
* Pacemaker,
* Emergency surgery and patients requiring rapid serial induction

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain with propofol injection | 5 minutes
  pain will be assessed using a four point behavioral scale: 1= no pain (no reaction); 2= mild pain (grimace); 3= moderate pain (grimace+cry); 4= severe pain (cry+withdrawal)

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)